CLINICAL TRIAL: NCT05062616
Title: Patient Satisfaction After Ingrown Toenail Surgery. A Review of 1200 Cases
Brief Title: Patient Satisfaction After Ingrown Toenail Surgery
Status: Completed | Type: Observational
Sponsor: Goztepe Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Esat UYGUR, Assoc.Prof.M.D., Goztepe Training and Research Hospital
Other Study IDs: 2021-03
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Ingrowing Nail With Infection
Keywords: patient satisfaction; operative treatment; ingrown toenail; onychocryptosis
MeSH Terms: conditions — Patient Satisfaction; Nails, Ingrown

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Toenail surgery — modified Winograd procedure

SUMMARY:
In this study, demographic characteristics (age, gender, which toe is involved, family history) of the patients who were operated because of ingrown nails were examined, and the post-operative satisfaction score of the patients was noted, and the recurrence rate and complications were recorded.

DETAILED DESCRIPTION:
The study was designed as single-center, single-surgeon observational study. Approximately 4000 patients who were operated on by the same surgeon between 2015-2020 due to ingrown nails were reached by phone, and patients' satisfaction was assessed by using the Surgical Satisfaction Questionnaire (SSQ-8). Outcomes such as retrospective treatment processes and complications were asked using a questionnaire, and patients' demographic characteristics were also recorded.

ELIGIBILITY:
Inclusion Criteria:

Patients who underwent ingrown toenail surgery Patients who could be reachable by phone over contact details on medical records

Exclusion Criteria:

Patients who were not reachable Patients who underwent another surgery on the targeted foot rather than ingrown toenail surgery Patients who had fractures on the targeted foot Clinical diagnosis of Alzheimer disease or patients who have lost their cognitive functions.

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had ingrown toenail surgery between 8 and 80 years old.
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
The Surgical Satisfaction Questionnaire (SSQ-8) | At least one year after surgery
  SSQ-8 is a validated tool for the assessment of patients who had been operated on.

SECONDARY OUTCOMES:
Recurrence | At least one year after surgery
  Recurrence rate is noted
The shape of nail clipping | through study completion, an average of 2 years
  straight or round cut
Family history | through study completion, an average of 2 years
  Positive or negatif family history

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Medeniyet University, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided